CLINICAL TRIAL: NCT07198633
Title: An Open-label, Multicenter Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-tumor Activity of QLC5508 and/or QLH12016 in Combination With Other Anti-tumor Therapies in Subjects With Advanced Prostate Cancer
Brief Title: A Clinical Study of QLC5508 and/or QLH12016 in Combination With Other Anti-tumor Therapies in Subjects With Advanced Prostate Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLC5508-202
Record Dates: First submitted 2025-09-15; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Advanced Prostate Cancer
MeSH Terms: interventions — Abiraterone Acetate; enzalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- QLC5508+NHA (Experimental)
  Interventions: Drug: QLC5508; Drug: abiraterone acetate; Drug: enzalutamide
- QLC5508+QLH12016 (Experimental)
  Interventions: Drug: QLC5508; Drug: QLH12016
- QLC5508+QLH12016+NHA (Experimental)
  Interventions: Drug: QLC5508; Drug: abiraterone acetate; Drug: enzalutamide; Drug: QLH12016
- QLH12016+NHA (Experimental)
  Interventions: Drug: QLC5508; Drug: abiraterone acetate; Drug: enzalutamide

INTERVENTIONS:
Drug: QLC5508 — B7H3 ADC; QLC5508 will be administered by injection at the dose and dosing frequency specified in the protocol.
Drug: abiraterone acetate — An oral CYP17 inhibitor; abiraterone acetate will be administered orally at the dose and dosing frequency specified in the protocol
  Arms: QLC5508+NHA; QLC5508+QLH12016+NHA; QLH12016+NHA
Drug: enzalutamide — An oral androgen receptor inhibitor; enzalutamide will be administered orally at the dose and dosing frequency specified in the protocol.
  Arms: QLC5508+NHA; QLC5508+QLH12016+NHA; QLH12016+NHA
Drug: QLH12016 — An oral androgen receptor PROTAC; QLH12016 will be administered orally at the dose and dosing frequency specified in the protocol
  Arms: QLC5508+QLH12016; QLC5508+QLH12016+NHA

SUMMARY:
This study is an open-label, multicenter Phase Ib/II clinical trial designed to evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-tumor activity of QLC5508 in combination with NHA (abiraterone or enzalutamide), QLC5508 in combination with QLH12016, QLC5508 in combination with QLH12016 and NHA (abiraterone or enzalutamide), and QLH12016 in combination with NHA (abiraterone or enzalutamide) in subjects with advanced prostate cancer.

The study consists of two stages:

Phase Ib: is the combination dose-escalation stage, during which the recommended Phase II dose (RP2D) will be determined.

Phase II is the efficacy exploration stage, in which, based on the RP2D established in Phase Ib, the therapeutic efficacy will be further evaluated in the target indication.

ELIGIBILITY:
Inclusion Criteria:

* The subject voluntarily agrees to participate and has signed the informed consent form.
* Male, aged ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
* Life expectancy of at least 3 months.
* Histologically or cytologically confirmed adenocarcinoma of the prostate.
* Radiologically confirmed metastatic prostate cancer.
* For subjects with mCRPC, serum testosterone must be at castrate levels, and they must have demonstrated either PSA progression or radiographic progression.
* Must have undergone surgical castration or be willing to receive medical castration.
* For Phase Ib, subjects must have experienced failure, intolerance, or refusal of standard therapy.
* Adequate function of major organs as defined by the protocol.
* Agreement to use effective contraception during the study (except for subjects who have undergone bilateral orchiectomy).
* Sufficient blood samples must be provided during the screening period for genetic mutation testing.

Exclusion Criteria:

* Prior treatment with the following agents: AR PROTAC, abiraterone, enzalutamide, or B7H3-targeted therapies.
* Presence of central nervous system (CNS) metastases, leptomeningeal metastases, or spinal cord compression requiring hormonal therapy.
* Receipt of extensive radiotherapy within 4 weeks prior to the first administration of the investigational medicinal product.
* Treatment with other investigational drugs or major surgery within 4 weeks prior to the first administration of the investigational medicinal product.
* Presence of factors that may affect drug administration, intake, or absorption.
* History of epilepsy, or a condition that could provoke seizures within 12 months prior to the first administration of the investigational medicinal product.
* Known history of substance abuse, alcoholism, or drug addiction; or prior history of significant neurological or psychiatric disorders, including dementia or hepatic encephalopathy.
* Presence of severe cardiovascular or cerebrovascular disease.
* Active, uncontrolled infection.
* Clinically uncontrolled third-space fluid accumulation prior to the first administration of the investigational medicinal product.
* History of other malignancies within 5 years prior to the first administration of the investigational medicinal product.
* Presence of moderate to severe pulmonary disease that significantly impairs lung function.
* For subjects receiving QLC5508, history of non-infectious interstitial lung disease (ILD) or pneumonitis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Phase Ib) | At the end of Day 28 after the first dose
  MTD is defined as the previous dose level at which 2 or more out of 2-6 subjects experienced a DLT
Maximum administered dose (MAD)(Phase Ib) | At the end of Day 28 after the first dose
  MAD is defined as follows: a) based on PK data, it is anticipated that at this dose level, the dose-exposure plateau has been reached, b) based on existing safety data, it is judged that dose escalation following this dose level will have a large safety risk or subject intolerance, or c) based on the PK-PD model, it suggested that the optimal target concentration of safety and efficacy has been explored.
recommended phase II dose (RP2D) (Phase Ib) | Through phase Ib completion, an average of 1 year.
  The RP2D will be comprehensively evaluated based on the safety, PK characteristics, and efficacy data from the Phase Ib study.
The incidence and severity of adverse events (AE) (Phase Ib) | Through phase Ib completion, an average of 1 year.
  Incidence and severity of adverse events (AEs) evaluated according to the NCI-CTCAE v5.0
PSA50 response（Phase II） | From Screening to confirmed progressive disease (approximately 1 year)
  Proportion of subjects with ≥ 50% PSA decrease
Objective response rate (ORR) (phase II) | From Screening to confirmed progressive disease (approximately 1 year)
  Best response until progression, as defined by RECIST 1.1 and PCGW3.